CLINICAL TRIAL: NCT07139535
Title: A Randomized, Double-blind, Placebo-Controlled Trial Comparing the Efficacy and Safety of RAY1225 Versus Placebo in Patients With Type 2 Diabetes, Inadequately Controlled With Diet and Exercise Alone
Brief Title: A Study of RAY1225 in Participants With Type 2 Diabetes Not Controlled With Diet and Exercise Alone
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAY1225-24-12
Record Dates: First submitted 2025-08-11; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: T2DM

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3mg RAY1225 (Experimental): Participants received 3 milligrams (mg) of RAY1225 as subcutaneous injection once every two week.
  Interventions: Drug: RAY1225
- 6mg RAY1225 (Experimental): Participants received 6 milligrams (mg) of RAY1225 as subcutaneous injection once every two week.
  Interventions: Drug: RAY1225
- 9mg RAY1225 (Experimental): Participants received 9 milligrams (mg) of RAY1225 as subcutaneous injection once every two week.
  Interventions: Drug: RAY1225
- Placebo (Placebo Comparator): Participants received placebo as subcutaneous injection once every two week.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: RAY1225 — Administered SC
  Arms: 3mg RAY1225; 6mg RAY1225; 9mg RAY1225
Drug: placebo — Administered SC
  Arms: Placebo

SUMMARY:
The goal for this study is to evaluate the efficacy and safety of RAY1225 versus placebo in participants with type 2 diabetes not under control with diet and exercise alone.

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed with type 2 diabetes mellitus (T2DM)
2. Having received only dietary and exercise therapy and never taken any antihyperglycemic medications before screening; OR Having taken no antihyperglycemic medications within the 12 weeks before screening and, prior to that, having received only oral antihyperglycemic drugs in a regimen of no more than two concomitant agents.
3. Have a body mass index (BMI) ≥20 kilograms per meter squared (kg/m²) at screening
4. Be of stable weight (±5%) for at least 12 weeks before screening

Exclusion Criteria:

1. Have type 1 diabetes mellitus
2. Presence of severe chronic diabetic complications at screening, including but not limited to: proliferative diabetic retinopathy, diabetic macular edema, and severe non-proliferative diabetic retinopathy requiring acute treatment;
3. History of diabetic ketoacidosis or hyperosmolar hyperglycemic state within 24 weeks prior to randomization;
4. Occurrence of a Grade 3 hypoglycemic event within 12 months prior to screening, or ≥3 Grade 2 hypoglycemic events (venous or capillary blood glucose <3.0 mmol/L) within 3 months prior to screening, or presence of hypoglycemia-related symptoms ;
5. History of severe trauma, severe infection, or surgery within 12 weeks prior to screening that may affect glycemic control;
6. Receipt of blood transfusion within 12 weeks prior to screening, or blood donation/loss ≥400 mL within 12 weeks prior to screening, or blood donation/loss ≥200 mL within 4 weeks prior to screening, or known hemoglobinopathy (such as thalassemia, hemolytic anemia, sickle cell anemia, etc.);
7. Any unstable or treatment-requiring endocrine disorders related to glycemic control other than type 2 diabetes mellitus (such as hyperthyroidism, acromegaly, Cushing's syndrome, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (HbA1c) | Baseline,36 Week
  HbA1c is the glycosylated fraction of hemoglobin A.

SECONDARY OUTCOMES:
Percentage of Participants Achieving an HbA1c Target Value of <7% | Baseline,36 Week
Percentage of Participants With HbA1c Target Value of <6.5% | Baseline,36 Week
Mean change in fasting serum glucose | Baseline,36 Week
Proportion of patients who achieved weight loss of >5%, >10%, and >15% from baseline | Baseline,36 Week

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijingcun, Hebei, China

IPD SHARING:
Plan to Share IPD: No